CLINICAL TRIAL: NCT00658294
Title: Analysis of the Potentially Parasitocidal Effect of a Long Term Chemotherapy With Benzimidazoles in Patients With Inoperable Alveolar Echinococcosis Using PET-CT and EmII/3-10 Serology
Brief Title: Analysis of the Potentially Parasitocidal Effect of a Long Term Chemotherapy With Benzimidazoles
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-1351
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Alveolar Echinococcosis
MeSH Terms: conditions — Alveolar echinococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Stop treatment

SUMMARY:
The aim of this study is to evaluate PET-CT and EmII/3-10 serology as potential markers to assess the parasitocidal effect of benzimidazoles

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Patients with inoperable alveolar echinococcosis
* With negative PET-CT
* EmII/3-10 serology under long-term chemotherapy with benzimidazoles

Exclusion criteria:

* Positive PET-CT
* Positive EmII-3-10 Serology
* No compliance
* Reduced life expectancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inoperable alveolar echinococchosis
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beat Müllhaupt 01 Studienregister MasterAdmins, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ammann RW, Stumpe KD, Grimm F, Deplazes P, Huber S, Bertogg K, Fischer DR, Mullhaupt B. Outcome after Discontinuing Long-Term Benzimidazole Treatment in 11 Patients with Non-resectable Alveolar Echinococcosis with Negative FDG-PET/CT and Anti-EmII/3-10 Serology. PLoS Negl Trop Dis. 2015 Sep 21;9(9):e0003964. doi: 10.1371/journal.pntd.0003964. eCollection 2015. PMID 26389799